CLINICAL TRIAL: NCT01703702
Title: A Randomized, Multicenter, Multicountry Study to Evaluate the Effectiveness of Florbetapir (18F) PET Imaging in Changing Patient Management and to Evaluate the Relationship Between Florbetapir (18F) PET Scan Status and Cognitive Decline
Brief Title: Effectiveness of Florbetapir (18F) PET Imaging in Changing Patient Management and the Relationship Between Scan Status and Cognitive Decline
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-A18
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Results first posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Subjects will receive florbetapir (18F) PET scans and physicians will have immediate access to PET scan results.
  Interventions: Drug: florbetapir (18F)
- Control (Experimental): Subjects will receive florbetapir (18F) PET scans but physicians will be blinded to PET scan results for 12 months
  Interventions: Drug: florbetapir (18F)

INTERVENTIONS:
Drug: florbetapir (18F) — Single i.v. bolus injection of 370MBq (10 mCi) followed by saline flush, 50 minutes prior to imaging, 10 minute image duration
  Other Names: 18F-AV-45; florbetapir F 18; AV-45; Amyvid

SUMMARY:
This study is designed to determine the effectiveness of florbetapir (18F) in changing patient management and to evaluate the association between scan status and cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

Patients may be enrolled in the mild impairment (not demented) group if the following criteria are met:

1. Males or females ≥ 50 to <= 90 years of age.
2. Have cognitive decline verified by a study partner or cognitive impairment verified by the study physician.
3. Have a study partner who provides separate consent and is willing to accompany the patient on all of the study visits.
4. Have an MMSE score of 24 to 30 inclusive.
5. Can tolerate a 10-minute PET scan.
6. Have the ability to cooperate and comply with all study procedures.
7. Have an enrolling physician who has less than high confidence in their diagnosis for the patient related to the cognitive decline at the time of enrollment.
8. Ability to provide informed consent for study procedures.

Patients may be enrolled in the dementia group if the following criteria are met:

1. Are males or females ≥ 50 to <= 90 years of age.
2. Meet clinical criteria for dementia.
3. Have a caregiver who provides separate consent and is willing to accompany the patient on all of the study visits.
4. Have an MMSE score of 16 to 24 inclusive.
5. Have not received a clinical examination and/or laboratory test results that strongly indicates a non-neurodegenerative cause for the patients cognitive impairment.
6. Can tolerate a 10-minute PET scan.
7. Have the ability to cooperate and comply with all study procedures.
8. Have an enrolling physician who has less than high confidence in their diagnosis for the patient related to the cognitive decline at the time of enrollment.
9. Ability to provide informed consent for study procedures. (If the patient is incapable of giving informed consent, the patient's legal representative may consent on behalf of the patient but the patient must still confirm assent. This person may serve as the study partner as well).

Exclusion Criteria:

Patients will be excluded from enrollment if they:

1. Have a current serious or unstable illness;
2. The patient or enrolling physician knows the result of a previous amyloid imaging scan;
3. The patient has a known brain lesion, pathology or alternative diagnosis that strongly explains the patient's clinical presentation;
4. Are receiving any investigational medications, or have participated in a trial with investigational medications within the last 30 days;
5. Have ever participated in an experimental study with an amyloid targeting agent (e.g. anti-amyloid immunotherapy, γ -secretase or β -secretase inhibitor) unless it can be documented that the patient received only placebo during the course of the trial;
6. Have had a radiopharmaceutical imaging or treatment procedure within 7 days prior to the study imaging session; or
7. Are females of childbearing potential who are not surgically sterile, not refraining from sexual activity or not using reliable methods of contraception.

Patients will also be excluded from enrollment if their enrolling physician:

1. Does not consider Alzheimer's disease as a potential cause of the patient's cognitive decline.
2. Is not the primary physician taking care of the patient with respect to the management of their cognitive impairment.
3. Cannot categorize the patient as either: a) having a documented and completed evaluation for cognitive decline within the past 18 months old; or b) currently undergoing evaluation for cognitive decline.
4. Is unwilling to suspend all testing and other evaluation procedures between the time of the baseline evaluation of the enrolling physician's diagnosis and management plan and the time the completion of the PET scan.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 2012-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (48):
- United States (18):
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Sun City, Arizona
  - Research Site, Clearwater, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Orlando, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Shreveport, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, Chestnut Hill, Massachusetts
  - Research Site, Quincy, Massachusetts
  - Research Site, Las Vegas, Nevada
  - Research Site, Patchogue, New York
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Providence, Rhode Island
  - Research Site, Salt Lake City, Utah
  - Research Site, Bennington, Vermont
- France (18):
  - Research Site, Amiens
  - Research Site, Bordeaux
  - Research Site, Bron
  - Research Site, Dijon
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nancy
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Reims
  - Research Site, Rouen
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Villeurbanne
- Italy (12):
  - Research Site, Bergamo
  - Research Site, Brescia
  - Research Site, Florence
  - Research Site, Genoa
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Monza
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Perugia
  - Research Site, Pisa
  - Research Site, Rome

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 641 patients enrolled in the study. 21 patients withdrew before receiving a florbetapir (F18) PET scan. 620 patients received florbetapir and comprise the Safety Population; 2 patients did not have a valid PET scan. Therefore; 618 patients were randomized to the intervention or control arms and comprise the Efficacy Population.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 308 | 310
Completed | 272 | 288
Not Completed | 36 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 308 | 310 | 618
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (8.2) | 72.7 (7.94) | 72.9 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 160 | 302
  Male | 166 | 150 | 316
Region of Enrollment [Number; unit: participants]
  United States | 112 | 111 | 223
  Italy | 109 | 112 | 221
  France | 87 | 87 | 174

OUTCOME MEASURES:

1. Primary Outcome: Clinical and Diagnostic Change in Patient Management
Description: Comparison of the percentage of patients who have a change in management from baseline to 3 months for patients who receive scan results immediately (intervention arm) and those who receive scan results 12 months later (control arm).
Time Frame: Baseline and 3 months
Population: Analysis population for this endpoint only includes those patients with both a baseline and follow-up value.
Measure: Number; unit: percentage of patients
Arm/Group | Intervention | Control
Number analyzed (Participants) | 300 | 299
percentage of patients | 68.0 | 55.5
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority or Other; p = 0.002, Chi-squared; Odds Ratio (OR) = 1.70, 95% CI 2-sided [1.22 to 2.38]

2. Primary Outcome: Change in ADAS-Cog 11 Total Score
Description: Change from baseline in the Alzheimer's Disease Assessment Scale - cognitive subscale (ADAS-cog) 11 Score in patients with mild impairment by positive or negative florbetapir (18F) PET scan result (Aß+/Aß-). ADAS-Cog scores (range 0-70) indicate performance on a series of 11 cognitive tasks where 0 indicates the highest level of cognitive performance and 70 indicates the lowest level of cognitive performance. Change in ADAS-Cog scores were calculated by subtracting the baseline score from the 12 month score. A change in ADAS-Cog greater than 0 indicates a deterioration in cognitive performance whereas a change in ADAS-Cog less than 0 indicates improved cognitive performance.
Time Frame: Baseline and 12 months
Population: Analysis population for this endpoint only includes those patients with mild cognitive impairment, and who reported both a baseline and follow-up value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Mild Impairment AB+: Patients diagnosed with a cognitive status of mild impairment and AB+ scan result.
- Mild Impairment AB-: Patients diagnosed with a cognitive status of mild impairment and AB- scan result.
Arm/Group | Mild Impairment AB+ | Mild Impairment AB-
Number analyzed (Participants) | 178 | 134
units on a scale | 0.95 (0.38) | 1.29 (0.43)
Statistical Analysis 1: Comparison: Mild Impairment AB+ vs Mild Impairment AB-; Test type: Superiority or Other; p = 0.568, ANCOVA; Adjusted for: Baseline ADAS-Cog score, study arm, Alzheimer's treatment, country, and interaction between study arm and Alzheimer's treatment; LS Mean Difference = -0.35, 95% CI 2-sided [-1.54 to 0.84]

3. Secondary Outcome: Change in Patient's Clinical Diagnosis
Description: Comparison of the percentage of patients who have a change in diagnosis from baseline to 3 months for patients in the intervention and control arms for whom the scan result was not predicted by the initial diagnosis.
Time Frame: Baseline and 3 months
Population: Analysis population for this endpoint only includes those patients whose scan result was not predicted by their baseline clinical diagnosis and recorded both a baseline and follow-up value.
Measure: Number; unit: percentage of patients
Groups:
- Intervention Scan/Diagnosis Discordant: Intervention arm patients whose florbetapir F18 PET scan results were not predicted by their baseline clinical diagnosis.
- Control Scan/Diagnosis Discordant: Intervention arm patients whose florbetapir F18 PET scan results were not predicted by their initial diagnosis
Arm/Group | Intervention Scan/Diagnosis Discordant | Control Scan/Diagnosis Discordant
Number analyzed (Participants) | 111 | 109
percentage of patients | 85.6 | 11.9
Statistical Analysis 1: Comparison: Intervention Scan/Diagnosis Discordant vs Control Scan/Diagnosis Discordant; Test type: Superiority or Other; p < 0.001, Chi-squared; Odds Ratio (OR) = 43.9, 95% CI 2-sided [20 to 96.12]

4. Secondary Outcome: Change in Diagnostic Confidence
Description: Comparison of the percentage point change in the physician's diagnostic confidence from baseline to month 3 in the intervention and control arms for patients whose scan result was predicted by their baseline clinical diagnosis. Diagnostic confidence was recorded by the physician as a whole number percent from 0-100% and the change in confidence was calculated by subtracting the baseline confidence from the confidence recorded at the specified timepoint. Values greater than zero reflect increased diagnostic confidence; values less than zero reflect decreased diagnostic confidence.
Time Frame: Baseline and 3 months
Population: Analysis population for this endpoint only includes those patients whose scan result was predicted by their baseline clinical diagnosis and recorded both a baseline and follow-up value.
Measure: Least Squares Mean (Standard Error); unit: Percentage Point
Groups:
- Intervention Scan/Diagnosis Concordant: Intervention arm patients whose florbetapir F18 PET scan results were predicted by their initial diagnosis
- Control Scan/Diagnosis Concordant: Control arm patients whose florbetapir F18 PET scan results were predicted by their initial diagnosis
Arm/Group | Intervention Scan/Diagnosis Concordant | Control Scan/Diagnosis Concordant
Number analyzed (Participants) | 189 | 190
Percentage Point | 23.54 (1.13) | 2.85 (1.15)
Statistical Analysis 1: Comparison: Intervention Scan/Diagnosis Concordant vs Control Scan/Diagnosis Concordant; Comparison of change in diagnostic confidence at follow-up (3 months); Test type: Superiority or Other; p < 0.001, ANCOVA; Adjusted for: Cognitive status (mild impairment/dementia), physician/practice type, country and florbetapir F18 PET scan result (Aß+/Aß-); LS Mean Difference = 20.69, 95% CI 2-sided [18.95 to 22.43]

5. Secondary Outcome: Change in Patient Management: Advice/Counseling
Description: Comparison of the percentage of patients in the intervention and control arms who have a change in management relating to advice and counseling from baseline to 3 months.
Time Frame: Baseline and 3 months
Population: Analysis population for this endpoint only includes those patients with both a baseline and follow-up value.
Measure: Number; unit: percentage of patients
Arm/Group | Intervention | Control
Number analyzed (Participants) | 300 | 299
percentage of patients | 64.7 | 58.9
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority or Other; p = 0.144, Chi-squared; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.92 to 1.78]

6. Secondary Outcome: Change in Caregiver Self-efficacy
Description: Comparison of the change in self-efficacy between intervention and control arms. Change in self-efficacy is defined as the difference between total score on the Fortinsky: Family caregivers' self-efficacy for managing dementia scale at Follow-up (3 months) and baseline. Self-efficacy for managing dementia is defined in terms of specific behaviors or tasks that can be learned, and that are highly relevant to daily management of the disease process. The scale consists of 10 questions, each with responses ranging from 1 (not at all certain) to 10 (very certain). The total score is calculated by summing the response for each item. The total score ranges from 10 to 100, with increasing scores representing increasing caregiver self-efficacy.
Time Frame: Baseline and 3 months
Population: Analysis population for this endpoint only includes those patients with both a baseline and follow-up value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 301 | 297
units on a scale | 0.16 (1.24) | 0.00 (1.26)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority or Other; p = 0.925, ANCOVA; Adjusted for: Baseline scale, Cognitive status (mild impairment/dementia), country and florbetapir F18 PET scan result (Aß+/Aß-); LS Mean Difference = 0.16, 95% CI 2-sided [-3.20 to 3.53]

7. Secondary Outcome: Change in Patient Management: Individual Categories
Description: Compare the percentage of patients with a change from baseline in the individual patient management categories at 3 months in the interventional and control arms.The individual categories are: Major diagnostic tests, Alzheimer's/cognition medication, neuropsychological tests, physician follow-up for re-evaluation or specialist referral.
Time Frame: Baseline and 3 months
Population: Analysis population for this endpoint only includes those patients with both a baseline and follow-up value.
Measure: Number; unit: percentage of patients
Arm/Group | Intervention | Control
Number analyzed (Participants) | 300 | 299
percentage of patients
  Major Diagnostic Tests | 21 | 20.4
  Alzheimer's/Cognitive Medication | 35.7 | 22.1
  Neuropsychological Tests | 14.7 | 9.7
  Physician Follow-up for Re-evaluation | 15.0 | 14.0
  Specialist Referral | 30.7 | 23.4
Statistical Analysis 1: Comparison: Intervention vs Control; Major Diagnostic Tests; Test type: Superiority or Other; p = 0.857, Chi-squared; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.70 to 1.54]
Statistical Analysis 2: Comparison: Intervention vs Control; Alzheimer's/Cognitive Medication; Test type: Superiority or Other; p < 0.001, Chi-squared; Odds Ratio (OR) = 1.96, 95% CI 2-sided [1.36 to 2.81]
Statistical Analysis 3: Comparison: Intervention vs Control; Neuropsychological Tests; Test type: Superiority or Other; p = 0.063, Chi-squared; Odds Ratio (OR) = 1.60, 95% CI 2-sided [0.97 to 2.64]
Statistical Analysis 4: Comparison: Intervention vs Control; Physician Follow-up for Re-evaluation; Test type: Superiority or Other; p = 0.741, Chi-squared; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.69 to 1.70]
Statistical Analysis 5: Comparison: Intervention vs Control; Specialist Referral; Test type: Superiority or Other; p = 0.046, Chi-squared; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.01 to 2.08]

ADVERSE EVENTS:
Time Frame: 48 hours post-injection
Groups:
- Safety Population: 620 patients received florbetapir (18F) and comprise the Safety Population.
Arm/Group | Safety Population
Serious Adverse Events (participants affected / at risk) | 2/620
Other Adverse Events (participants affected / at risk) | 36/620
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=620)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=620)
Flushing (Vascular disorders) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 17 (17)
Dizziness (Nervous system disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Asthenia (General disorders) | 3 (3)
Fatigue (General disorders) | 3 (3)
Feeling abnormal (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Hallicination, olfactory (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Abnormal faeces (Gastrointestinal disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less